CLINICAL TRIAL: NCT00929877
Title: A Randomised Double Blind, Placebo-controlled, Parallel-group Study of the Efficacy and Safety of 2 Doses of Ketoprofen Lysinate Lozenges (6.25 mg & 12.5 mg) in Patients With Sore Throat
Brief Title: KRYSTAL- KetopRofen lYsinate Sore ThroAt Lozenges
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KETOP_C_03968; 2008-008265-36(EudraCT)
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Ketoprofen lysinate 12.5 mg (Experimental)
  Interventions: Drug: KETOPROFEN(RP19583)
- Ketoprofen lysinate 6.25 mg (Experimental)
  Interventions: Drug: KETOPROFEN(RP19583)
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KETOPROFEN(RP19583) — Oral administration up to a maximum of 5 lozenges within a 24-hour period during 3 days
  Arms: Ketoprofen lysinate 12.5 mg
Drug: KETOPROFEN(RP19583) — Oral administration up to a maximum of 5 lozenges within a 24-hour period during 3 days
  Arms: Ketoprofen lysinate 6.25 mg
Drug: Placebo — Oral administration up to a maximum of 5 lozenges within a 24-hour period during 3 days
  Arms: Matching placebo

SUMMARY:
Primary Objective:

To compare the single-dose efficacy of ketoprofen lysinate lozenges (6.25 mg and 12.5 mg ketoprofen base) with placebo, on total pain relief summed over 15 to 120 min (TOTPAR15-120) after the first intake of study drug.

Secondary Objectives:

To compare the single-dose efficacy of ketoprofen lysinate lozenges (6.25mg and 12.5mg ) with placebo after the first intake on:

* the total pain relief summed over 15 to 360min (TOTPAR15-360)
* the changes from baseline of global throat pain intensity assessed over 15 to 120min and over 15 to 360min.
* the changes from baseline of throat soreness over 15 to 120min and over 15 to 360min
* the changes from baseline of swollen throat over 15 to 120min and over 15 to 360min To compare pain relief, global throat pain intensity, throat soreness and swollen throat in the evening of days 1, 2 and 3

To evaluate the safety of ketoprofen lysinate lozenges (6.25mg and 12.5mg ) and placebo at follow-up visit on:

Day 4: - adverse events and clinical examination Day 7: - adverse events reporting (followed by a clinical examination if needed)

ELIGIBILITY:
Inclusion criteria:

* Patients with a sore throat associated or not with an URTI > or = 24 hours and < or = 6 days' duration, in the absence of A.Streptococcus*,
* Evidence of tonsillo-pharyngitis (TPA score > or = 5) at inclusion,
* With a score of throat soreness > or = 6 (0-10 ordinal scale),
* With a perception of swollen throat > or = 60mm (VAS),
* With a global throat pain intensity such as pain at swallowing
* assessed by a VAS > or = 60 mm.

  *Specific exploration at Inclusion:
* The Score of Mac Isaac will be performed by the investigator.
* Presence of streptococcus will be assessed by a throat swab test Patients having a positive swab test will not be included.

Exclusion criteria:

* Patients having used any local medication containing a local oral anesthetic such as lozenge, spray, mouth rinse or any topical throat treatment within 2 hours before study entry
* Patients with positive throat swab test for A.Streptococcus pharyngitis
* Patients having used analgesics within 4 hours before study entry
* Patients having used any long-acting or slow release analgesics within 12 hours before study entry
* Patients having used any anti inflammatory treatment 8-12 hours before study entry
* Patients having used any anti histaminic 8-12 hours before study entry
* Patients with pharyngeal paresthesia
* Patients with pharyngeal mycosis
* Patients with known history of ketoprofen, aspirin or other NSAID-induced bronchospasm
* Hypersensitivity to ketoprofen or its excipients
* Any disease that could compromise breathing such as bronchopneumonia or asthma
* Evidence of mouth-breathing or uncomfortable coughing
* Any chronic disease that requires a long period anti-inflammatory treatment
* Any chronic disease that requires long term use of anticoagulants or use of anticoagulants or anti-platelet agents one week before study entry,
* Women known to be pregnant.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The TOTPAR15-120 which is the sum of each pain relief scale score | measured every 15 minutes during the 2 hours following the first study drug intake

SECONDARY OUTCOMES:
The TOTPAR15-360 which is the sum of each pain relief scale score | Measured every 15 minutes during the 2 hours following the first study drug intake at study site then every hour up to 6 hours as outpatient.
The global throat pain intensity | assessed every 15 min during 2 hours after the first study drug intake
The morning pain relief scale score | measured in morning of days 1, 2 and 3
The evening pain relief scale score | measured in evening of days 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Perdriset, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Frankfurt, Germany
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Barcelona, Spain